CLINICAL TRIAL: NCT00153114
Title: PolyethyleneGlycol3350 Laxative vs Placebo in Constipated Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 851-15
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

INTERVENTIONS:
Drug: polyethyleneglycol3350

SUMMARY:
Assess the safety and efficacy of polyethyleneglycol3350 laxative as compared to placebo therapy in pediatric patients with a history of constipation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients between the ages of 4 to 16 years.
* Adolescent female patients must not be pregnant or lactating.
* constipated according to ROME I definition
* Two or fewer bowel movements during the initial observation week.
* Absence of a stool impaction
* Bowel movement after receiving enema
* Are otherwise in good health, as judged by a physical examination.
* Parent or guardian is mentally competent to sign an instrument of informed consent

Exclusion Criteria:

* Patients with heme positive stool at baseline exam.
* Patients with fecal impaction at baseline, or after the observation period, as indicated by physical exam
* Patients with known or suspected perforation or obstruction other than fecal impaction.
* Patients who are breastfeeding, pregnant or intend to become pregnant during the study.
* Female patients of childbearing potential who refuse a pregnancy test.
* Patients with a known history of organic cause for their constipation.
* Patients with congenital malformations that produce constipation (Hirschsprung's disease, imperforate anus, children with cerebral palsy or other neurologic abnormalities, or systemic diseases).
* History of gastric retention, inflammatory bowel disease, bowel resection, or colostomy.
* Use of concomitant medications that cause constipation
* Patients who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Patients with known allergy to polyethyleneglycol or polyethyleneglycol containing medications.
* Patients with clinically significant elevations of TSH or abnormal plasma electrolytes.
* Patients who, within the past 30 days have participated in an investigational clinical study

Ages: 4 Years to 16 Years | Sex: All
Age Groups: Child
Enrollment: 100
Dates: Start 2003-01; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Greater than 2 bowel movements per week

SECONDARY OUTCOMES:
Analysis of individual ROME I criteria
Safety (adverse event and laboratory testing)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Nurko, MD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Boston, Massachusetts
  - Morristown, New Jersey
  - Pittsburgh, Pennsylvania